CLINICAL TRIAL: NCT01447199
Title: The Molecular Predisposition to Hereditary Nonpolyposis Colon Cancer (HNPCC)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: DM94-060
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Bladder Cancer; Colorectal Cancer; Endometrial Cancer; Kidney Cancer; Skin Cancer; Uterus Cancer
Keywords: Bladder cancer; Colorectal cancer; Endometrial cancer; Kidney cancer; Skin cancer; Uterus cancer; Molecular Predisposition; Hereditary Nonpolyposis Colon Cancer; HNPCC; Molecular genetic testing; Gene mutations; Mutation analyses; Genetic polymorphisms; Family history of cancer; Early age of cancer onset; Little/no personal or family history of cancer; Spouses; Questionnaires; Blood sample; Saliva Sample
MeSH Terms: conditions — Urinary Bladder Neoplasms; Colorectal Neoplasms; Endometrial Neoplasms; Kidney Neoplasms; Skin Neoplasms; Uterine Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Health; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will have a single sample (8-10 teaspoons) of blood collected at M. D. Anderson, depending upon current health status. In the case of individuals not coming to the clinic, a blood drawing kit will be sent to the participant's home, which will include instructions and a postage-paid return express mail envelope. If participant unable or unwilling to give a blood sample, saliva samples can be collected instead.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Gene Mutation: Group with increased risk for developing colorectal and/or other cancers as the result of an inherited gene mutation, family history of cancer, or an early age of cancer onset.
  Interventions: Behavioral: Health and Diet Questionnaire
- No Cancer History: Group with little/no personal or family history of cancer.
  Interventions: Behavioral: Health and Diet Questionnaire
- Spouses: Spouses of those who may have an increased risk for developing colorectal and/or other cancers as the result of an inherited gene mutation, family history of cancer, or an early age of cancer onset, or little/no personal or family history of cancer.
  Interventions: Behavioral: Health and Diet Questionnaire

INTERVENTIONS:
Behavioral: Health and Diet Questionnaire — Mailed questionnaires asking about foods eaten, cooking methods as well as overall health, and vitamin/medication use, taking several hours to complete.
  Other Names: Survey

SUMMARY:
The goal of this study is to understand factors which may influence risk for colorectal and other cancers in families. These factors include genetic variability, in combination with diet and lifestyle. In order to achieve these goals, we need to contact as many eligible participants as possible.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will have a single sample (8-10 teaspoons) of blood collected, depending upon current health status. The blood will be drawn at MD Anderson. If you cannot come to the clinic, a blood drawing kit will be sent to the your home, which will include instructions and a postage-paid return express mail envelope. Phlebotomy charges connected to this study will be paid by the study. The blood sample will be sent to a research laboratory at MD Anderson for analyses. If you are unwilling or unable to give a blood sample, you can give a saliva sample instead. In this case, a kit will be mailed to you with instructions for obtaining the saliva sample. A prepaid envelope will be included for its return. Participants who previously participated in Protocol PA11-0567 and provided a blood sample do not need to provide another blood sample. The previously stored blood sample collected by Protocol PA11-0567 may be used.

You will be asked to answer a series of questions. These questions will ask about foods eaten either one year ago or one year before the first diagnosis of cancer. There will also be questions about cooking methods as well as overall health, and vitamin and medication use. Some of the questions are personal, but all answers will be kept strictly private.

The questionnaire will be sent to your home via U.S. or express mail. It may take several hours to complete the survey, but there is no time limit on its completion. There are no right or wrong answers to the questions. A postage-paid return envelope will be provided for the return of the questionnaire.

Solid tumor material and colonoscopy specimens of normal tissue will be collected from participants requiring either colonoscopy or surgery for routine clinical reasons. The tumor fragments will be collected from specimens. Tissue required for a clinical pathology diagnosis will not be used for research purposes.

This is an investigational study. About 2,000 patients and family members will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with a new referral for a diagnosis of colorectal cancer (adenocarcinoma) and/or HNPCC-related cancers at the UTMDACC will be considered potentially eligible for this study regardless of prior treatment.
2. Families maintained at the UTMDACC Hereditary Colon Cancer Registry that have a known germline mutation in a mismatch repair gene or contain two or more first degree relatives diagnosed with CRC and/or any HNPCC-related cancers, one of whom must be less than or equal to 50 years at diagnosis.
3. First-degree and more distant relatives of individuals diagnosed with CRC and/or any HNPCC-related cancers from either of the groups in 1 and 2 (above).
4. Any patient diagnosed with CRC and/or any HNPCC-related cancers less than or equal to 45 years of age.
5. Greater than or equal to age 18 at time of study.
6. Able to provide informed consent to participate in this study indicating that they are aware of the investigational nature, in keeping with the policies of this hospital.
7. Non-HNPCC quartets, defined as parents and two offspring who do not carry a mismatch repair gene mutation. These non-HNPCC quartets should have no personal history of cancer, nor cancer in any first degree relatives of the quartet members, nor history of trinucleotide repeat syndromes. Non-HNPCC parents in a quartet should be less than 34 years old at the time the offspring were born.
8. Lynch Syndrome patients identified and recruited through Protocol PA11-0567 who opt into Optional Procedure B, which consents the patient to participate in this study.

Exclusion Criteria:

1. Diagnosis of current major psychiatric disorder, per DSM-III-R (or DSM IV).
2. Age less than 18 years at time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Referrals from Departments of GI Oncology, GI Medicine and Nutrition, GI Surgery, GYN Oncology, Cancer Prevention and from the Genetic Counselors at UT MD Anderson Cancer Center, families and spouses.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 1994-09 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Time to Onset for Colorectal Cancer | Overall study period up to 15 years.
  Primary endpoint is time to onset for colorectal cancer using Cox proportional hazard regression for determining the role that polymorphic variants of genes have on risk for development of HNPCC at an early age.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Lynch, MD, JD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org